CLINICAL TRIAL: NCT01499732
Title: An Exploratory Trial to Evaluate Premature Endothelial Dysfunction, as Measured by Positron Emission Tomography (PET) Scan With Cold Pressor Test (CPT), in Patients With Early Rheumatoid Arthritis (RA) Compared to Patients With Established RA, and Normal Subjects. Additionally, the Relationship Between the PET Scan Findings and the Inflammatory, Cardiovascular Risk, and Endothelial Dysfunction Biomarkers Will be Analyzed
Brief Title: Exploratory Trial to Evaluate Premature Endothelial Dysfunction in Early Rheumatoid Arthritis(RA)Compared to Patients With Established RA, and Normal Subjects
Status: Completed | Type: Observational
Sponsor: Orrin M Troum, M.D. and Medical Associates (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-320
Record Dates: First submitted 2011-12-15; First posted 2011-12-26 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Premature Endothelial Dysfunction; Rheumatoid Arthritis; Healthy
Keywords: Premature endothelial dysfunction; Early Rheumatoid Arthritis; established rheumatoid arthritis; Premature endothelial dysfunction in early rheumatoid arthritis; Premature endothelial dysfunction in established rheumatoid arthritis; Endothelial function in healthy subjects
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Early Rheumatoid Arthritis: Subjects currently experiencing active early rheumatoid arthritis (duration of symptoms < or = 2 years) according to the 2010 ACR/EULAR criteria for the diagnosis of RA at screening. Must be drug naive (no prior treatment with traditional disease-modifying antirrheumatic drugs (DMARDs), or biologic response modifying agents)
- Healthy subjects without rheumatoid arthritis: Healthy subjects without rheumatoid arthritis
- Established Rheumatoid Arthritis: Subjects currently experiencing active established rheumatoid arthritis (duration fo symptoms > or = 2 years) according to the 2010 ACR/EULAR criteria at screening. Subjects with active established RA currently receiving methotrexate, must have received it for at least 12 weeks, and at a stable dose (> or = 15 mg/week) for at least 6 weeks prior to screening. They must be biologic naive, and must recieve at least 5mg oral folic acid weekly

SUMMARY:
Premature Endothelial Dysfunction is present in patients with early rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

Group 1

1. Subjects currently experiencing active early RA (duration of symptoms ≤ 2 years) according to the 2010 ACR/EULAR criteria for the diagnosis of RA at screening.
2. Subjects with early RA must be drug naïve (no prior treatment with traditional disease-modifying antirheumatic drugs (DMARDs), or biologic response modifying agents).

   Group 2
3. Subjects currently experiencing active established RA (duration of symptoms ≥ 2 years) according to the 2010 ACR/EULAR criteria for the diagnosis of RA at screening.
4. Subjects with active established RA currently receiving methotrexate (MTX), must have received it for at least 12 weeks, and at a stable dose (≥15mg/week) for at least 6 weeks prior to screening. They must be biologic drug naïve. These subjects must receive at least 5 mg oral folic acid weekly.
5. Subjects diagnosed with RA must be seropositive with documented rheumatoid factor (RF) or anti-cyclic citrullinated peptide (anti CCP) positivity. If a documented history of RF or anti CCP positivity is not available, RF and anti CCP titers will be obtained at screening Group 3
6. Healthy subjects without RA.
7. All subjects must have sitting diastolic BP ≤90 mm Hg and/or sitting systolic BP ≤ 140 at screening
8. Subjects must have fasting plasma glucose (FPG) of ≤ 100 mg/dL.
9. If subjects with established RA are receiving an oral corticosteroid, the dose must be ≤7 mg/day prednisone (or equivalent) and stable for at least 28 days prior to screening.
10. Subjects able and willing to give written informed consent and comply with the requirements of the study protocol. Informed consent must be obtained prior to any study-related procedures.

    A copy of the signed informed consent form must be given to the subject
11. Patients must have a BMI of less than 42

Exclusion Criteria:

1. Major surgery (including joint surgery) within 8 weeks prior to screening.
2. Rheumatic autoimmune disease other than RA, including systemic lupus erythematosus (SLE), mixed connective tissue disease (MCTD), scleroderma, polymyositis, or significant systemic involvement secondary to RA (vasculitis, pulmonary fibrosis or Felty's syndrome). Prior history of or current inflammatory joint disease other than RA (gout, Lyme disease, seronegative spondyloarthropathy including reactive arthritis and psoriatic arthritis)
3. Functional class IV as defined by ACR Classification of Functional Status in RA
4. Current treatment with any traditional DMARDs other than MTX within 4 weeks before the screening visit (For subjects with established RA). Current or prior use of Leflunomide will be exclusionary.
5. Treatment with any investigational agent within 4 weeks (or 5 half-lives of investigational agent, whichever is longer) before screening
6. Exposure to any Biologic Response Modifying Agent for RA
7. Intraarticular or parenteral corticosteroids within 6 weeks prior to screening (For subjects with established RA)
8. Exclusionary laboratory: Serum creatinine >2 mg/dL, ALT or AST > 2.0 x ULN, total bilirubin > 2.0 x ULN, platelet count <100 x 10⁹ /L, hemoglobin < 8.5 g/dL, WBC count < 1,000/mm³ , absolute neutrophil count < 1,000/ mm³, absolute lymphocyte count < 500/mm³, triglycerides >400 mg/dL, Serum potassium <3.5 or >5.5 mEq /L without medication, serum albumin <2.5 g/dL, Gamma GT 3.0 x UNL
9. Smokers (use of tobacco products in the recent past < 6 months). Urine cotinine levels will be measured during screening for all subjects. Smokers will be defined as any subject who reports cigarette use or has a urine cotinine greater than 200 ng/mL.
10. Pregnant women or nursing mothers
11. Females of child bearing potential who are not using reliable means of contraception
12. Evidence of serious uncontrolled concomitant cardiovascular (including known CAD, HTN, or hyperlipidemia), nervous system, pulmonary, renal, hepatic, endocrine or GI disease.
13. Uncontrolled disease states, such as asthma, psoriasis, or inflammatory bowel syndrome, where flares are commonly treated with corticosteroids.
14. History or presence of severe bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated).
15. History of cardiovascular abnormalities including myocardial infarction, angina pectoris, hypertensive encephalopathy, stroke, transient ischemic attack, valvular heart disease, ventricular arrhythmia A-V block, atrial fibrillation or cardiac revascularization/angioplasty. Symptoms or clinical evidence of congestive heart failure or known left ventricular ejection fraction < 40%.
16. Medical history of clinically significant ECG abnormalities, including history of a prolonged QT-interval syndrome.
17. History of autonomic dysfunction
18. Known active current or history of recurrent bacterial, viral, fungal, mycobacterial, or other infections such as atypical mycobacterial disease, hepatitis B and C, HIV, herpes zoster, or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening.
19. Any malignancy except for skin cancer (basal cell or squamous cell) diagnosed within the previous 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Five adults (>18 years of age), male or non pregnant, non nursing female with active early rheumatoid arthritis (<2 years), five adults, male or non-pregnant, non nursing female with active established rheumatoid arthritis (>2 years), and five healthy adults, male or non-pregnant, non nursing female without RA are to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To evalute the presence of endothelial dysfunction in patients with rheumatoid arthritis utilizing PET/CT scan with cold pressor test. | 5 months
  Endothelial dysfunction will be defined as myocardial blood flow (MBF)during cold pressor test (CPT)of less than or equal to 40%

SECONDARY OUTCOMES:
To evaluate the relationship between PET Scan findings and biomarkers (inflammatory, cardiovascular risk and endothelial dysfunction), and outcome measures | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Orrin M Troum, MD, Principal Investigator — Orrin M. Troum, MD and Medical Associates
Locations (1):
- Orrin M. Troum, MD and Medical Associates, Santa Monica, California, United States